CLINICAL TRIAL: NCT06020079
Title: The Effect of Laughter Yoga on Depressıon and Serotonın Levels ın Patients Who Have Been Patıent Wıth Bariatric Surgery
Brief Title: Laughter Yoga Effect Depression, Serotonin Levels With Bariatric Surgery Patient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tokat Gaziosmanpasa University (Other)
Collaborators: Inonu University (Other)
Responsible Party: Principal Investigator, Gulnaz Kizilkaya, Assistant profesör, phD, Tokat Gaziosmanpasa University
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Supportive Care
Other Study IDs: InonuU
Record Dates: First submitted 2023-08-22; First posted 2023-08-31 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Bariatric Surgery; Depression
Keywords: bariatric surgery; depression; laughter yoga; nursing; serotonin
MeSH Terms: conditions — Depression | interventions — Laughter Therapy

STUDY DESIGN:
Intervention Model Description: A Guasi-experimental Study with a Pretest-Posttest Control Group Design.
Who Masked: Participant
Masking Description: who had undergone bariatric surgery in the general surgery ward of the university hospital 6-24 months ago. Sample size was determined using power analysis. The analysis revealed that the sample should consist of a total of 62 patients (31 intervention, 31 control),
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- laughter yoga group (Experimental): Laughter yoga was administered to the intervention group twice a week, on Tuesdays and Fridays, for 5 weeks, in a total of 10 sessions (the duration of each session was 50 minutes). Apart from the first and last sessions, eight sessions of the laughter yoga intervention were held via an Internet program with on-line meeting option due to the COVID-19 pandemic that started in March 2019. For the feasibility of online sessions, opinions were obtained from experts who provide laughter yoga leadership training.
  Interventions: Other: laughter yoga
- Control group (No Intervention): no intervation

INTERVENTIONS:
Other: laughter yoga — According to the literature and the training received on laughter yoga, the time required for the treatment of depression is 50 minutes. The first 10 minutes includes relaxation, stretching and warm-up exercises. The next 30 minutes includes laughing exercises, and finally, the last 10 minutes includes relaxation exercises.
  Steps of laughter yoga sessions:
  1. Clapping hands and warm-up exercises: Participants clap their hands, fingers and palms. Then, sounds like ho-ho and ha-ha are added to the clapping exercises along with the rhythm.
  2. Deep breathing exercises: Breathing exercises should be repeated 3-4 times while standing
  3. Childlike games: Arms are raised, imitating the funny and clumsy behavior of a child.
  4. Laughter exercises: The researcher names the exercise, explains how to do it, and the group performs the exercise together.
  Dance and Relaxation
  Arms: laughter yoga group

SUMMARY:
The goal of this a quasi-trial model with pre and post-test control group is to determine the effect of laughter yoga on depression and serotonin levels in patients undergoing bariatric surgery.

The main question's it aims to answer are:

* Question 1: Does laughter yoga reduce the level of depression in patients undergoing bariatric surgery?
* Question 2: Does laughter yoga increase serotonin levels in patients who have undergone bariatric surgery? 158 patients who underwent bariatric surgery in the General Surgery Service of a university hospital in Malatya/Turkey and 6-24 months after the operation participated in the study. Sample size was determined using power analysis and 62 patients were sampled. 31 patients were determined as the control group and 31 patients as the experimental group. 10 sessions of laughter yoga were applied to the patients in the experimental group who agreed to participate in the study that met the criteria. No intervention was made in the control group.

DETAILED DESCRIPTION:
The first stage of the data, identifying the patients, was collected by the researcher in the general surgery service of the hospital determined between February-June 2021.The patient information and blood samples, which are the second phase of the data, were collected by the researcher at the same time intervals in the nursing faculty meeting room of the designated university. In order to determine the participants to participate in the research, the participants who met the criteria were contacted by phone and an appointment was requested. Face-to-face Beck Depression Scale was applied to the patients who attended the appointment in the General Surgery service. 158 patients who got 17 points from the Beck Depression Scale were determined among the 62 patients who agreed to participate in the study, the first 31 experimental groups and the second 31 control groups. Before their hospital visit for the interview, the patients were reminded that they should be fasting for blood sample collection and they should be on a 24-hour serotonin free diet. All participants filled the Patient Information Form as a pre-test in the nursing faculty meeting room and gave blood samples for serotonin levels. Laughter yoga was applied to the experimental group twice a week, on Tuesdays and Fridays, for 2,5 months, for a total of 10 sessions (each session 50 minutes) by the researcher after obtaining a laughter yoga practice certificate. Due to the COVID-19 pandemic that started during this study period, the first and last sessions were applied face-to-face, and the other eight sessions of laughter yoga were carried out with an internet program that allows online meetings. Expert opinions from laughter yoga leaders for online applicability of laughter yoga taked. After 10 sessions were applied to the participants, the Beck Depression Scale was re-administered to the participants in the experimental group as a post-test and blood samples were taken again to check the serotonin levels. The Beck Depression Scale was re-administered 5 weeks after the pretest without any intervention in the control group, and blood samples were taken again to determine serotonin levels.

ELIGIBILITY:
Inclusion Criteria:

* Residing in the city where the research was conducted
* Having received a score of 17 or higher on the Beck Depression Scale
* Not receiving any psychological treatment
* Having no communication problems

Exclusion Criteria:

* Having consumed foods containing serotonin (banana, walnut, tomato, eggplant, hazelnut, peanut, avocado, pineapple, kiwi, melon, dairy products, fish, eggs) in the last 24 hours on the days of blood collection
* Having diseases that may cause physical strain and increase intra-abdominal pressure during laughter yoga (e.g., bleeding hemorrhoids, all kinds of hernia, persistent cough, severe back pain, heart diseases, high blood pressure, urinary incontinence, epilepsy, complications of late morbid obesity such as anastomotic leakage, extreme nausea-vomiting, dumping syndrome, and reflux).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Measured by the Beck Depression Scale that laughter yoga would reduce depression | 2,5 months
  The scale was developed by Beck et al. in 1961. Hisli conducted the Turkish validity and reliability studies of the scale in 1989 . The scale consists of 21 items assessing the symptoms that develop during depression. While the lowest score of the scale is 0, the highest score is 63. Scores between 5 and 9 indicate normal depression; scores between 10-18 indicate mild-moderate depression; scores between 19-29 indicate moderate-severe depression; and scores between 30-63 indicate severe depression. High scores indicate higher levels of depression. The cut-off point of the scale is 17. The reliability analysis of the scale showed that the Cronbach's alpha coefficient is 0.80. In our study, the pre-test Cronbach α of the Beck Depression Scale was calculated as 0.628, while the post-test Cronbach α was calculated as 0.841.
It was measured by the ELISA method by experts in the laboratory environment that laughter yoga would increase serotonin levels. | 2,5 months
  Before taking blood from the patients, they were asked whether they fasted and followed a 24-hour serotonin-restricted diet. Approximately 6 ml of venous blood samples were taken from the participants with 10 ml injectors and placed into yellow- and red-capped blood collection tubes. The blood samples were centrifuged in the laboratory of the physiology department of the medical faculty of a university. The serum part of the centrifuged blood was placed in godets and kept in the -45 degree-refrigerators until all the blood was collected. Labels containing the patients' names, surnames and dates were attached to the godets. All frozen serums and kits were then allowed to reach room temperature for 15 minutes and processed using the ELISA method. DRG (serotonin fast elisa EIA-5061) brand kits were worked on in accordance with the package insert. The detection range of the kits was 10.2-2500 ng/ml and the sensitivity was 6.2 ng/ml.

CONTACTS AND LOCATIONS:
Overall Officials: meral özkan, phD, Principal Investigator — thessis advisor
Locations (1):
- inonuU, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: national thesis center — http://161.9.164.68/xmlui/handle/11616/61878